CLINICAL TRIAL: NCT00621387
Title: Double-Blind, Placebo-Controlled Study of Three-Month Treatment With the Combination of Ofloxacin and Roxithromycin in Recent-Onset Reactive Arthritis
Brief Title: Study of Long-Term Antibiotic Treatment in Reactive Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 121-853-93
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2007-11

CONDITIONS: Reactive Arthritis
Keywords: reactive arthritis; antibiotics
MeSH Terms: conditions — Arthritis, Reactive | interventions — Ofloxacin; Roxithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ofloxacin and roxithromycin
  Interventions: Drug: ofloxacin and roxithromycin
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ofloxacin and roxithromycin — 150 mg roxithromycin tablet twice daily and 200mg ofloxacin tablet twice daily for 3 months
  Other Names: Tarivid and Surlid
  Arms: 1
Drug: placebo — placebo tablets identical to ofloxacin and roxithromycin twice daily for 3 months
  Arms: 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial of the effect of 3-month treatment with the combination of 200 mg ofloxacin twice daily and 150 mg roxithromycin twice daily on clinical course of recent-onset reactive arthritis. Patients are followed-up at regular intervals until 6 months. The main outcome measure is recovery from arthritis, and secondary outcome measures include swollen and tender joint counts, Ritchie index, joint pain, serum C-reactive protein level and blood erythrocyte sedimentation rate. The study will also address the safety and tolerability of long-term antibiotic treatment. 56 patients are enrolled and the enrollment of patients has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute reactive arthritis
2. Preceding infection confirmed by positive culture and/or serology, or with a history of urethritis or gastroenteritis within the preceding 2 months
3. Age 18 or older

Exclusion Criteria:

1. Allergy to quinolones or macrolides
2. Treatment with systemic corticosteroids within 2 weeks
3. Serum creatinine level elevated over the reference limit
4. Alanine aminotransferase or alkaline phosphatase levels elevated over twice the reference limit
5. Current or planned pregnancy, or lack of contraception
6. Known HIV positivity
7. Blood leukocyte count less than 4.0x109/l
8. Blood platelet count less than 100x109/l
9. Lack of co-operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1993-11; Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients recovered from arthritis | 6 months

SECONDARY OUTCOMES:
Swollen joint count | 6 months
Tender joint count | 6 months
Ritchie index | 6 months
Joint pain (visual analogue scale) | 6 months
Serum C-reactive protein level | 6 months
Blood erythrocyte sedimentation rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marjatta Leirisalo-Repo, MD, Principal Investigator — Division of Rheumatology, Department of Medicine, Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Division of Rheumatology, Department of Medicine, Helsinki
  - Peijas Hospital, Vantaa